CLINICAL TRIAL: NCT00092599
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Efficacy, Safety, and Tolerability of Ezetimibe 10 mg or Placebo Co-administered With Existing Simvastatin 10 mg or 20 mg in Attaining Low-Density Lipoprotein Cholesterol Target Levels in Patients With Hypercholesterolemia and Coronary Heart Disease.
Brief Title: Investigational Drug Study in Patients With Elevated Cholesterol and Coronary Heart Disease (0653-801)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-801; 2004_039
Record Dates: First submitted 2004-09-23; First posted 2004-09-27 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Coronary Disease
Keywords: Elevated Cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653, ezetimibe
Drug: Comparator: ezetimibe, placebo

SUMMARY:
This study will evaluate patients who have coronary heart disease to determine if an investigational drug will further lower cholesterol when taken in combination with an approved cholesterol lowering medication.

DETAILED DESCRIPTION:
The duration of treatment is 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elevated cholesterol and coronary heart disease

Exclusion Criteria:

* Patients who do not meet specific cholesterol levels as required by the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2003-02; Primary Completion 2004-06 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching LDL goal of <2.60 mmol/L after 6 weeks of treatment

SECONDARY OUTCOMES:
Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Brohet C, Banai S, Alings AM, Massaad R, Davies MJ, Allen C. LDL-C goal attainment with the addition of ezetimibe to ongoing simvastatin treatment in coronary heart disease patients with hypercholesterolemia. Curr Med Res Opin. 2005 Apr;21(4):571-8. doi: 10.1185/030079905X382004. PMID 15899106